CLINICAL TRIAL: NCT00548847
Title: A Pilot Phase II Study of Immunotherapy for the Treatment of AML, ALL, BP CML, and MDS Relapsed After Allogeneic Transplantation
Brief Title: Immunotherapy for Acute Myeloid Leukemia (AML), Acute Lymphoblastic Leukemia (ALL), Blast Phase Chronic Myelogenous Leukemia (BP CML), and Myelodysplastic Syndrome (MDS) Relapse After Allogeneic Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Martha Arellano, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002219; WCI1228-06 (Other: Winship Cancer Institute of Emory University)
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Leukemia
Keywords: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Introns; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GM-CSF, Interferon-α-2b (Experimental)
  Interventions: Biological: GM-CSF; Biological: Interferon-α-2b

INTERVENTIONS:
Biological: GM-CSF — Dosing schedule: 250 mcg/m² subcutaneously Mon-Wed-Fri. Response assessed between 2 and 4 weeks. Duration on study is 3 months.
  Other Names: Sargramostim; Leukine; Rhu GM-CSF; NSC #617589
Biological: Interferon-α-2b — Dosing schedule: 1.5 mcg/kg subcutaneously Monday weekly. Response assessed between 2 and 4 weeks. Duration on study is 3 months.
  Other Names: Interferon-alpha-2b; Intron A®; Pegylated Interferon-α-2b; Peg-Intron; Peginterferon alfa-2b

SUMMARY:
The relapse of acute leukemia, MDS and blast phase CML after allogeneic transplantation affects approximately 1/3 to 1/2 of all transplant recipients and is the main cause of treatment failure. There is currently no effective standard treatment for this condition.

This study will test the activity and feasibility of using a regimen to boost the immune system in order to treat AML, ALL, blast phase CML, and MDS relapse after allogeneic transplantation.

DETAILED DESCRIPTION:
This is a pilot phase II open label study testing the activity and feasibility of utilizing a regimen to boost the immune system in order to treat AML, ALL, blast phase CML, and MDS relapse after allogeneic transplantation. The regimen is a step-wise use of withdrawal of immunosuppression, cytoreduction if needed, administration of granulocyte-macrophage colony-stimulating factor (GM-CSF) and pegylated interferon (IFN) α-2b to patients who relapsed after an allogeneic transplant and will assess efficacy.

Relapse is the major problem following allogeneic hematopoietic progenitor cell transplants. There is currently no standard way to treat leukemia that relapsed after transplant, and patients have a poor prognosis.

A retrospective analysis of patients treated at Emory showed that administration of GM-CSF and interferon-alpha-2b was well-tolerated and affected long-term remissions in a small number of relapsed patients (after allogeneic transplant). Pre-clinical and clinical data from ours and other centers showed that relapsed leukemic blasts have down-regulation of co-stimulatory molecules and a tendency to evade the immune system. Cytokines can up-regulate co-stimulatory molecules on leukemic blasts and have been shown to increase the cytotoxicity of T-cells. This effect may be beneficial as a graft vs. leukemia effect for patients with relapse after allogeneic transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 1 year.
2. Patients who have received an allogeneic transplant to treat AML, ALL, MDS, or CML and have relapse or progression of their AML, ALL, MDS, or CML are eligible to participate in the study. Relapse is defined as: reappearance of leukemic blasts as determined by morphologic analysis of the blood or marrow, reappearance of a phenotypic population of leukemia blasts by flow cytometric analysis of the blood or marrow, reappearance of a chromosome abnormality which is associated with the original leukemia as determined by chromosomal or fluorescence in situ hybridization (FISH) testing (ex: a translocation between chromosomes 9 and 22 for CML), reappearance of the molecular marker which is associated with the original leukemia as determined by polymerase chain reaction (PCR) (ex: breakpoint cluster region [BCR]-Abelson murine leukemia [ABL] for CML or ALL).

   *Patients who received allogeneic transplantation to treat AML, ALL, MDS, or CML with detectable disease, and did not achieve remission of their leukemia after transplant are eligible.
3. Eastern Cooperative Oncology Group (ECOG) performance status < 2 for adults, and Lansky status 60% for children.
4. Liver functions tests (aspartate transaminase [AST]/alanine aminotransferase [ALT]/bilirubin) < 5x the upper limit of normal.
5. Creatinine < 3x the upper limit of normal.
6. Lack of active grade 2-4 acute graft-versus-host disease (GVHD) 3 weeks after discontinuation of immunosuppression.
7. Patients with limited stage and extensive stage chronic GVHD of mild severity (lichenoid changes), or requiring < prednisone 10 mg/m² daily will be included.
8. Recipients of grafts procured from related and unrelated donors with any level of human leukocyte antigen (HLA)-matching.

Exclusion Criteria:

1. Pregnant patients are excluded due to unknown risk to the unborn fetus with cytokines.
2. Allergy to components of interferon-alpha-2b or GM-CSF.
3. Current uncontrolled infection.
4. Current grade 2-4 acute GVHD or chronic extensive GVHD of moderate to severe nature, requiring treatment with more than 10 mg/m² of prednisone daily.
5. Uncompensated heart failure, New York Heart Association (NYHA) class III-IV:

   * Class I: patients with no limitation of activities; they suffer no symptoms from ordinary activities;
   * Class II: patients with slight, mild limitation of activity; they are comfortable with rest or with mild exertion;
   * Class III: patients with marked limitation of activity; they are comfortable only at rest;
   * Class IV: patients who should be at complete rest, confined to bed or chair; any physical activity brings on discomfort and symptoms occur at rest.
6. Breast feeding, due to unknown risk to the infant.
7. Inability to give informed consent.
8. Children under 1 year of age.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Arellano, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were enrolled at the Winship Cancer Institute of Emory University. The study closed to accrual in May 2011.
Groups:
- GM-CSF, Interferon-α-2b: Granulocyte-macrophage colony-stimulating factor (GM-CSF), Interferon-α-2b: Dosing schedule: GM-CSF, 250 mcg/m2 Mon-Wed-Fri; Pegylated Interferon-α-2b 1.5 mcg/kg Monday weekly. Response assessed between 2 and 4 weeks. Duration on study is 3 months.
Period: Overall Study
Arm/Group | GM-CSF, Interferon-α-2b
Started | 15
Completed | 8
Not Completed | 7
Not completed — Disease progression | 7

BASELINE CHARACTERISTICS:
Groups:
- GM-CSF, Interferon-α-2b: GM-CSF, Interferon-α-2b: Dosing schedule: GM-CSF, 250 mcg/m2 Mon-Wed-Fri; Pegylated Interferon-α-2b 1.5 mcg/kg Monday weekly. Response assessed between 2 and 4 weeks. Duration on study is 3 months.
Arm/Group | GM-CSF, Interferon-α-2b
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 13
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of GM-CSF and Pegylated Interferon-alpha 2b When Administered to Patients With AML, ALL, Blast Phase CML, and MDS Relapse After Allogeneic Transplantation, Defined as Progression-free Survival of > 33% at 3 Months
Description: Efficacy is defined as progression-free survival of > 33% at 3 months. This is based on our retrospective data on 10% 3 month survival for relapsed patients. Progression is defined an an increase in blasts in blood or marrow by 50% compared to baseline with at least 20% of all cells being blasts at the time of assessment.
Time Frame: 3 months after cytokine treatment
Measure: Number; unit: percentage of progression-free patients
Groups:
- GM-CSF, Interferon-α-2b: GM-CSF, Interferon-α-2b: Dosing schedule: GM-CSF, 250 mcg/m² Mon-Wed-Fri; Pegylated Interferon-α-2b 1.5 mcg/kg Monday weekly. Response assessed between 2 and 4 weeks. Duration on study is 3 months.
Arm/Group | GM-CSF, Interferon-α-2b
Number analyzed (Participants) | 15
percentage of progression-free patients | 13

2. Secondary Outcome: Overall Survival at 6 Months (Evaluate Overall Responses; Perform Lab Experiments to Test Hypothesis That Exposure to Interferon-alpha and GM-CSF Up-regulates Co-stimulatory Molecule Expression on Relapsed Acute Leukemia Cells)
Time Frame: 6 months after cytokine treatment
Measure: Number; unit: participants
Arm/Group | GM-CSF, Interferon-α-2b
Number analyzed (Participants) | 15
participants | 2

ADVERSE EVENTS:
Arm/Group | GM-CSF, Interferon-α-2b
Serious Adverse Events (participants affected / at risk) | 8/15
Other Adverse Events (participants affected / at risk) | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF, Interferon-α-2b (N=15)
Death (General disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Infection (Infections and infestations) | 2
Hemorrhage (Blood and lymphatic system disorders) | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF, Interferon-α-2b (N=15)
Fever (General disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Malaise (General disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Nausea (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes